CLINICAL TRIAL: NCT03897127
Title: Randomized Phase III Study of Standard Intensive Chemotherapy Versus Intensive Chemotherapy With CPX-351 in Adult Patients With Newly Diagnosed AML and Intermediate- or Adverse Genetics
Brief Title: Study of Standard Intensive Chemotherapy Versus Intensive Chemotherapy With CPX-351 in Adult Patients With Newly Diagnosed AML and Intermediate- or Adverse Genetics
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Ulm (Other)
Collaborators: Jazz Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Verena Gaidzik, Principal Investigator, University of Ulm
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AMLSG 30-18
Record Dates: First submitted 2019-03-19; First posted 2019-04-01 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Acute Myeloid Leukemia
Keywords: CPX-351; Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Cytarabine; Daunorubicin; CPX-351

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard arm (Active Comparator)
  Interventions: Drug: Cytarabine; Drug: Daunorubicin
- Investigational arm (Experimental)
  Interventions: Drug: CPX-351

INTERVENTIONS:
Drug: Cytarabine — Induction therapy: 200 mg/m2 i.v. (continuously) d1-7
  Consolidation therapy:
  * Patients age 18-60 years
    o Intermediate-dose cytarabine 1500 mg/m2 i.v. q12h (3 hrs) d1-3
  * Patients age >60 years o Intermediate-dose cytarabine 1000 mg/m2 i.v. q12h (3 hrs) d1-3
  Arms: Standard arm
Drug: Daunorubicin — Induction therapy: 60 mg/m2 i.v. (1 hr) d1-3
  Arms: Standard arm
Drug: CPX-351 — Induction 1:
  o CPX-351 44 mg/m2 daunorubicin / 100 mg/m2 cytarabine [100 U/m²] i.v. (90 min) d1,3,5
  Induction 2:
  o CPX-351 44 mg/m2 daunorubicin / 100 mg/m2 cytarabine [100 U/m²] i.v. (90 min) d1,3
  Consolidation therapy:
  o CPX-351 29 mg/m2 daunorubicin / 65 mg/m2 cytarabine [65 U/m²] i.v. (90 min) d1,3
  Arms: Investigational arm

SUMMARY:
The trial is a randomized, open-label phase III study comparing CPX-351 vs conventional intensive induction and consolidation chemotherapy in patients with newly diagnosed AML and intermediate- or adverse-risk genetics (according to 2017 ELN criteria), including AML with myelodysplasia-related changes (AML-MRC) and therapy-related AML according to the World Health Organization (WHO) classification. Overall survival (OS) in the restricted set of de novo patients will be the primary endpoint.

ELIGIBILITY:
Patient Inclusion Criteria:

1. Patients with newly diagnosed AML and intermediate- or adverse-risk genetics (according to 2017 ELN criteria [Appendix B]), including AML with myelodysplasia-related changes (AML-MRC) and therapy-related AML according to the World Health Organization (WHO) classification
2. Age ≥ 18 years, no upper age limit
3. Patient considered eligible for intensive chemotherapy
4. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2 at screening
5. Genetic assessment in AMLSG central laboratory
6. Adequate renal function as evidenced by serum creatinine ≤ 2.0 × ULN or creatinine clearance >40 mL/min based on the Cockcroft-Gault glomerular filtration rate (GFR)
7. Adequate hepatic function as evidenced by:

   * Serum total bilirubin ≤ 1.5 × upper limit of normal (ULN) unless considered due to Gilbert's disease, or leukemic involvement following approval by the Coordinating Investigator or Co-Coordinating Investigator
   * Aspartate aminotransferase (AST), alanine aminotransferase (ALT), and alkaline phosphatase (ALP) ≤ 3.0 × ULN, unless considered due to leukemic involvement following approval by the Coordinating Investigator or Co-Coordinating Investigator
8. No prior chemotherapy for acute leukemia except hydroxyurea for up to 14 days during the diagnostic screening phase for the control of peripheral leukemic blasts in patients with leukocytosis (e.g., white blood cell [WBC] counts >30x109/l); prior treatment of myelo-dysplastic syndrome with hypomethylating agents is allowed
9. Non-pregnant and non-nursing women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test within a sensitivity of at least 25 mIU/mL within 72 hours prior to randomization ("Women of childbearing potential" is defined as a sexually active mature woman who has not undergone a hysterectomy or bilateral oophorectomy or who has had menses at any time in the preceding 24 consecutive months)
10. Female patients of childbearing potential must agree to avoid getting pregnant while on therapy and for 27 weeks after the last dose of study drug
11. Women of childbearing potential must either commit to continued abstinence from heterosexual intercourse or apply one highly effective method of birth control (such as IUD, bilateral tubal ligation, or partner's vasectomy) in combination with one acceptable method of birth control at the same time (such as hormonal contraception or the male partner has to use a latex condom coated with spermicide lubricant or combined with spermicide gel or foam) while on therapy and for 27 weeks after the last dose of study drug. Hormonal contraception is only a highly effective method of birth control in case of combined (estrogen and progestogen containing) associated with inhibition of ovulation or progestogen-only hormonal contraception associated with inhibition of ovulation is used
12. Men must use a latex condom coated with a spermicide lubricant or combined with spermicide gel or foam during any sexual contact with women of childbearing potential, even if they have undergone a successful vasectomy and must agree to avoid to father a child (while on therapy and for 6 months after the last dose of study drug). In addition, their female partners of childbearing potential have to use a highly effective method of birth control
13. Able to understand and willing to sign an informed consent form (ICF)

Patient Exclusion Criteria:

1. AML with favorable-risk genetics according to 2017 ELN criteria [Appendix B]:

   * AML with t(8;21)(q22;q22.1), RUNX1-RUNX1T1
   * AML with inv(16)(p13.1q22)/t(16;16)(p13.1;q22), CBFB-MYH11
   * AML with mutated NPM1 without FLT3-ITD or with FLT3-ITDlow
   * AML with biallelic CEBPA mutation
2. AML with FLT3 mutation as assessed by DNA fragment analysis PCR for FLT3-ITD and FLT3-TKD mutation. Positivity is defined as a FLT3-ITD or FLT3-TKD / FLT3-WT ratio of ≥ 0.05 (5%).
3. Acute promyelocytic leukemia (APL) with t(15;17)(q22;q12); PML-RARA; or one of the other pathognomonic variant chromosomal translocations/ fusion genes
4. AML with BCR-ABL1
5. Prior treatment of myelodysplastic syndrome (MDS) with intensive chemotherapy or bone marrow transplant with a curative intent
6. Significant active cardiac disease within 6 months prior to the start of study treatment, including New York Heart Association (NYHA) class III or IV congestive heart failure; myocardial infarction, unstable angina and/or stroke; severe cardiac arrhythmias, or left ventricular ejection fraction (LVEF) <50% by ultrasound obtained within 28 days prior to the start of study treatment
7. Severe obstructive or restrictive ventilation disorder
8. Uncontrolled infection
9. Clinical symptoms suggestive of active central nervous system (CNS) leukemia or known CNS leukemia. Evaluation of cerebrospinal fluid (CSF) during screening is only required, if there is a clinical suspicion of CNS involvement by leukemia during screening
10. Evidence of active hepatitis B or C infection or known Human Immunodeficiency Virus (HIV) infection
11. Patients with a "currently active" second malignancy. Patients are not considered to have a currently active malignancy, if they have completed therapy and are considered by their physician to be at < 30% risk of relapse within one year. However, subjects with the following history/concurrent conditions are allowed:

    * Basal or squamous cell carcinoma of the skin
    * Carcinoma in situ of the cervix
    * Carcinoma in situ of the breast
    * Incidental histologic finding of prostate cancer
12. Severe neurological or psychiatric disorder interfering with ability to give an informed consent
13. No consent for registration, storage and processing of the individual disease characteristics and course as well as information of the family physician about study participation
14. No consent for biobanking of patient's biological specimens
15. Current participation in any other interventional clinical trial within 30 days before the first administration of the investigational product or at any time during the trial
16. Patients with prior cumulative anthracycline exposure of daunorubicin (or equivalent) can be included but the maximum of daunorubicin (or equivalent) dose of 550 mg/m2 must not be exceeded. Anthracycline-based therapy should be avoided until exposure to the previous cardiotoxic agents is negligible. If this is not possible, the patient's cardiac function should be carefully monitored and an absolute cumulative dose of 400 mg/m² in adults can be exceeded only with great caution. In patients who received radiation therapy to the mediastinum the maximum of daunorubicin (or equivalent) dose of 400 mg/m2 must not be exceeded.
17. Known or suspected hypersensitivity to cytarabine, daunorubicin or liposomal products and/or any excipients
18. History of Wilson's disease or other copper-metabolism disorder
19. Receipt of live, attenuated vaccine within 30 days prior to the inclusion in the clinical trial (NOTE: Subjects, if enrolled, should not receive live vaccine during the trial and until 6 months after the therapy).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 882 (Estimated)
Dates: Start 2019-09-04 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) in the restricted set of de novo patients | 2 years

SECONDARY OUTCOMES:
Overall survival (OS) in the extended set of patients | 2 years
Event-free survival (EFS) with CRi considered as response to induction therapy in both, the restricted set of de novo patients and the extended set of patients | 2 years
Event-free survival (EFS) with CRi considered as failure of induction therapy in the restricted set of de novo patients | 2 years
Rate of objective response in the restricted set of de novo patients | 2 months
  complete remission [CR], CR with incomplete hematologic recovery [CRi], CRi without measurable residual disease [CRiMRD-], CR without measurable residual disease [CRMRD-])

OTHER OUTCOMES:
EFS with CRi considered as failure of induction therapy in the extended set of patients | 2 years
  Exploratory endpoint
Response rates (CR/CRi/CRMRD-/CRiMRD-) in the extended set of patients | 2 years
  Exploratory endpoint
Relapse-free survival (RFS) in patients who achieved CR/CRi during induction chemotherapy | 2 years
  Exploratory endpoint
Relapse-free survival (RFS) in patients who achieved CR during induction chemotherapy | 2 years
  Exploratory endpoint
Cumulative incidence of relapse (CIR) in patients who achieved CR/CRi during induction chemotherapy | 2 years
  Exploratory endpoint
Cumulative incidence of relapse (CIR) in patients who achieved CR during induction chemotherapy | 2 years
  Exploratory endpoint
Cumulative incidence of death (CID) in patients who achieved CR/CRi during induction chemotherapy | 2 years
  Exploratory endpoint
Cumulative incidence of death (CID) in patients who achieved CR during induction chemotherapy | 2 years
  Exploratory endpoint
EFS with allogeneic HCT considered as competing event | 2 years
  Exploratory endpoint
RFS with allogeneic HCT considered as competing event | 2 years
  Exploratory endpoint
CIR with allogeneic HCT considered as competing event | 2 years
  Exploratory endpoint
CID with allogeneic HCT considered as competing event | 2 years
  Exploratory endpoint
OS with allogeneic HCT considered as competing event | 2 years
  Exploratory endpoint
QoL NCI PRO-CTCAE (National Cancer Institute) Patient Reported Outcomes Common Terminology Criteria for Adverse Events questionnaire) | 2 years
  PRO-CTCAE responses are scored from 0 to 4, whereas lower values represent a better outcome. For this trial, the burden of symptoms that will be captured by this questionnaire comprises nausea, diarrhea, rash, and alopecia.
QoL EORTC QLQ-FA12 | 2 years
  The EORTC QLQ-FA12 module complements the core EORTC QLQ-C30 questionnaire regarding fatigue. . Each item can be scored in four dimension on a scale from 1 to 4 with higher scores indicating worse symptoms.
QoL EORTC QLQ-C30 (Core Quality of Life Questionnaire developed by European Organization for Research and Treatment of Cancer) | 2 years
  The EORTC QLQ-C30 subscale scores are transformed to a 0 to 100 scale, with higher scores on functional scales indicating better function and higher scores on symptom scales indicating worse symptoms.
Rate of hospitalization including admissions at intensive care unit (ICU) | 8 months
  Exploratory endpoint
Reasons for hospitalization | 8 months
  Exploratory endpoint
days of hospitalization by treatment setting | 8 months
  Exploratory endpoint
rate of use of anti-infectives and other medications, e.g. against nausea or vomiting | 8 months
  Exploratory endpoint
additional therapies administered | 8 months
  Exploratory endpoint
place of chemotherapy administration (inpatient vs outpatient setting) | 8 months
  Exploratory endpoint
duration of administration | 8 months
  Exploratory endpoint
number of outpatient visits | 8 months
  Exploratory endpoint
Frequency of salvage therapies | 8 months
  Exploratory endpoint
Incidence and intensity of adverse events (AEs) according to Common Terminology Criteria for Adverse Events (CTCAE) version v5.0 | 2 years

CONTACTS AND LOCATIONS:
Locations (62):
- Austria (6):
  - Medizinische Universität Graz, Graz
  - Tirol Kliniken GmbH Innsbruck, Innsbruck
  - Ordensklinikum Linz GmbH, Elisabethinen, Linz
  - Feldkirch, Landeskrankenhaus, Rankweil
  - Landeskrankenhaus Salzburg, Salzburg
  - Hanuschkrankenhaus Wien, Vienna
- Germany (56):
  - Klinikum Aschaffenburg, Aschaffenburg
  - Helios Klinikum Bad Saarow, Bad Saarow
  - Berlin Charite - Campus Charite Mitte, Berlin
  - Vivantes Klinikum Am Urban, Berlin
  - Berlin Charite - Campus Benjamin Franklin, Berlin
  - Vivantes Klinikum Neukölln, Berlin
  - Charité Berlin, Berlin
  - Bochum, Augusta-Kranken-Anstalt, Bochum
  - Knappschaftskrankenhaus Bochum-Langendreer, Bochum
  - Universitätsklinikum Bonn, Bonn
  - Städtisches Klinikum Braunschweig gGmbH, Braunschweig
  - Klinikum Bremen-Mitte, Bremen
  - Klinikum Darmstadt, Darmstadt
  - St.-Johannes-Hospital, Dortmund
  - Universitätsklinikum Düsseldorf, Düsseldorf
  - Kliniken Essen Süd, Ev. Krankenhaus Essen- Werden gGmbH, Essen
  - Klinikum Esslingen, Esslingen am Neckar
  - Malteser Krankenhaus St. Franziskus-Hospital, Flensburg
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Universitätsklinikum Gießen, Giessen
  - Katholisches Karl-Leisner-Klinikum gGmbH, Wilhelm-Anton-Hospital gGmbH Goch, Goch
  - Universitätsmedizin Greifswald, Greifswald
  - Asklepios Kliniken Hamburg GmbH St. Georg, Hamburg
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Asklepios Klinik Altona, Hamburg
  - Evangelisches Krankenhaus Hamm gGmbH, Hamm
  - Klinikum Region Hannover - Klinikum Siloah, Hanover
  - Medizinische Hochschule Hannover, Hanover
  - SLK-Kliniken GmbH Heilbronn, Heilbronn
  - Marienhospital Herne, Klinikum der Ruhr, Herne
  - Kaiserslautern, Westpfalz-Klinikum, Kaiserslautern
  - Städtisches Klinikum Karlsruhe gGmbH, Karlsruhe
  - Klinikum Lippe-Lemgo, Lemgo
  - Klinikum der Stadt Ludwigshafen am Rhein gGmbH, Ludwigshafen
  - Universitätsklinikum Schleswig-Holstein, Lübeck
  - Klinikum Lüdenscheid, Lüdenscheid
  - Universitätsklinikum Magdeburg, Magdeburg
  - Klinikum der Johannes Gutenberg Universität, Mainz
  - Klniikum Hochsauerland GmbH, Meschede
  - Johannes Wesling Klinikum Minden, Minden
  - Klinikum rechts der Isar München, München
  - Ortenau Klinikum, Offenburg-Gengenbach, Offenburg
  - Pius Hospital Oldenburg, Oldenburg
  - Klinikum Oldenburg AöR, Oldenburg
  - Klinikum Passau, Passau
  - Universitätsklinikum Regensburg, Regensburg
  - Marienhaus Klinikum St. Elisabeth Saarlouis, Saarlouis
  - Klinikum Stuttgart, Stuttgart
  - Stuttgart, Diakonie-Klinikum, Stuttgart
  - Klinikum Traunstein, Traunstein
  - Mutterhaus der Borromäerinnen, Trier
  - Krankenhaus der Barmherzigen Brüder Trier, Trier
  - Universitätsklinikum Tübingen, Tübingen
  - Universitätsklinikum Ulm, Ulm
  - Schwarzwald-Baar Klinikum Villingen- Schwenningen GmbH, Villingen-Schwenningen
  - Helios Klinikum Wuppertal, Wuppertal